CLINICAL TRIAL: NCT01429935
Title: Comparison of The Anti Inflammatory and Analgesic Effect of Ginger and Ibuprofen in Post Surgical Pain Model; a Randomized,Placebo-controlled,Double-blind Clinical Trial
Brief Title: Anti Inflammatory and Analgesic Effect of Ginger Powder in Dental Pain Model
Acronym: GPE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, farshid rayati, assisstant proffessor of oral and maxillofacial department, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 504
Record Dates: First submitted 2011-09-04; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Impacted Third Molar Tooth
Keywords: dental pain model; Ginger powder; CRP
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ginger powder (Active Comparator)
  Interventions: Drug: Ginger powder
- Ibuprofen (Active Comparator): capsules of Ibuprofen 400 mg
  Interventions: Drug: Ibuprofen
- placebo (Placebo Comparator): capsules contain starch
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Ginger powder — capsules contain 500mg Ginger powder,every 6hours,for 5 days
  Other Names: zintoma
  Arms: Ginger powder
Drug: Ibuprofen — capsules of Ibuprofen 400 mg, every 6 hours for 5 days
  Arms: Ibuprofen
Other: placebo — capsules contain starch
  Arms: placebo

SUMMARY:
Ginger contains constituents with pharmacological properties similar to the novel class of dual-acting NSAIDs. Compounds in this class inhibit arachidonic acid metabolism via the cyclooxygenase (COX) and lipooxygenase (LOX) pathways. These compounds have notably fewer side effects than conventional NSAIDs and now are being investigated as a novel class of anti-inflammatory compounds. Although ginger has potentially strong anti-inflammatory components, its efficacy on acute inflammation was not assessed before. The common postoperative sequelae of surgical removal of impacted teeth are pain, trismus and swelling, related to local inflammatory reaction, with cyclooxygenase and prostaglandins playing a crucial role. NSAIDs (e.g. Ibuprofen) are effective in the management of postoperative dental pain, likely through blockage of prostaglandin synthesis and are commonly used. The efficacy of Ibuprofen in the treatment of postoperative dental pain has been evaluated in several clinical trials. However, NSAIDs are contraindicated in patients with gastrointestinal ulcers, bleeding disorders, and renal dysfunctions. Therefore, there is a need for an effective, oral analgesic with a more favorable safety profile. The primary aim of this study was to investigate the ability of Ginger powder (Zintoma, Goldaru) to reduce postoperative swelling, pain and trismus in an acute pain model.

DETAILED DESCRIPTION:
Ginger, the rhizome of Zingiber officinale, has a long history of medicinal use. In traditional Chinese and Indian medicine, ginger has been used to treat a wide range of ailments including stomachache, diarrhea, nausea, asthma, respiratory disorders, toothache, gingivitis, and arthritis. Subsequent studies revealed that ginger contains constituents with pharmacological properties similar to the novel class of dual-acting NSAIDs. Compounds in this class inhibit arachidonic acid metabolism via the cyclooxygenase (COX) and lipooxygenase (LOX) pathways. These compounds have notably fewer side effects than conventional NSAIDs and now are being investigated as a novel class of anti-inflammatory compounds. Different animal studies revealed that oral dried ginger or ginger extract reduced inflammation in paw and joint swelling induced by different chemical agents, lung inflammation induced by lipopolysaccharides (LPS) and arthritis induced by collagen . Several clinical studies support the value of ginger for the treatment of osteoarthritis . In addition to alleviating pain, ginger extract has been reported to decrease joint swelling. In some of these trials it was reported that ginger relieved pain and swelling to varying degrees in patients with osteoarthritis and rheumatoid arthritis as well as those with muscular pain without causing any adverse effects during a period ranging from 3 months to 2.5 years . In one recent trial ginger was tested in primary dysmenorrhea in comparison with Ibuprofen and mefenamic acid and no significant differences was found between the three study groups in relief, stability, or aggravation of symptoms . The common postoperative sequelae of surgical removal of impacted teeth are pain, trismus and swelling, related to local inflammatory reaction, with cyclooxygenase and prostaglandins playing a crucial role. NSAIDs (e.g. Ibuprofen) are effective in the management of postoperative dental pain, likely through blockage of prostaglandin synthesis and are commonly used. The efficacy of Ibuprofen in the treatment of postoperative dental pain has been evaluated in several clinical trials . However, NSAIDs are contraindicated in patients with gastrointestinal ulcers, bleeding disorders, and renal dysfunctions. Therefore, there is a need for an effective, oral analgesic with a more favorable safety profile. The primary aim of this study was to investigate the ability of Ginger powder (Zintoma, Goldaru,Iran) to reduce postoperative swelling, pain and trismus after third molar surgery.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one mesio-angular impacted mandibular third molar(5-7 difficulty degree)
* adults without any kind of systemic disease
* adults with at least Diploma educational degree

Exclusion Criteria:

* history of cold,fever,infection or any other inflammatory conditions during one month before surgery
* known allergy to NSAIDs ,ginger or acetaminophen
* any kind of hematopoietic or bleeding disorders
* pregnancy or lactating
* history of peptic ulceration
* history of corticosteroid use
* duration of surgery more than 30 minutes
* any infection, fever or any kind of disease cause on days 1,2 and 3 after surgery
* failure to attend for follow up
* using any kind of medication other than given drugs until day 5 post operatively
* being on anticoagulants except for mini-aspirin (72-325 mg/day)
* mentally incapable of understanding or complying with the study protocol or for failing to sign the informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Decreased amount of cheek swelling after surgery | 5 days
  Using standard calipers, cheek thickness will be measured from the lingual aspect of the mid-portion of the crown of the mandibular 1st molar (on the same side) to the tangent of the skin of the cheek.

SECONDARY OUTCOMES:
Decreased amount of serum CRP levels | 3 days
  A venous blood sample (approximately 4 ml, 2ml for CBC check up and 2 ml for CRP concentration) will be collected to quantitatively assess the CRP concentration after surgery and the second sample will be collected 72 hours postoperatively
Amount of pain severity | 5 days
  using 100mmVAS scale,at 1 hour intervals in the first 12 hours following the surgery and every 6 hours until day 5.
Increased amount of Mouth opening ability | 5 days
  assessed by measuring the distance between the upper and lower central incisal edges at maximal mouth opening on days 0 (baseline) and 1,3 and 5 post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Farshid Rayati, DDS,OMFS, Study Chair — Assisstant professor of oral and maxillofacial dapartment; Fateme Hajmanuchehri, Study Director — Assisstant professor of general pathology department; Mehran Purghasemi, Study Director — General pharmacologist; Elnaz Najafi, DDS, Study Director — General dentist; Farshid Rayati, DDS,OMFS, Principal Investigator — Assisstant professor of oral and maxillofacial department; Elanaz Najafi, dentist, Principal Investigator — General dentist
Locations (2):
- Iran (2):
  - Qazvin University of Medical Sciences, Qazvin, Qazvin State
  - University of Medical Science, Qazvin